CLINICAL TRIAL: NCT06970340
Title: Pilot Program: Effect of "Online MedEd" Intern Bootcamp Training on First Year Residents' Well-being and Skills Confidence. A Randomized Controlled Trial
Brief Title: Online MedEd Intern Bootcamp: Hybrid (Online+Live) Training for First Year Residents
Acronym: 2024-OME-RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Raji Ayinla, Director of Medicine, New York City Health and Hospitals Corporation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-08-221
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Burnout Among First Year Residents
Keywords: Interns; Bootcamp; Burnout; Wellness; First Year Resident
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Crossover timeline:
  First group July 15 2024 - January 05 2025 Second group January 06 2025 - June 15 2025
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Enrolled into a 6-month online training program plus biweekly live discussion sessions from July 15 2024 to January 15 2025
  Interventions: Behavioral: Online MedEd Intern Bootcamp
- Control (No Intervention): Residency training as usual. No access to online training platform or live sessions.

INTERVENTIONS:
Behavioral: Online MedEd Intern Bootcamp — 6 months of online access plus biweekly live sessions
  Arms: Intervention

SUMMARY:
This study is testing a web-based "Intern Boot Camp" from Online MedEd to see if it can make the first year of residency less stressful for new internal-medicine doctors at Harlem Hospital. Right after orientation, residents are randomly placed into one of two groups:

Intervention group - gets six months of free access to the Bootcamp videos plus twice-a-week, one-hour review sessions led by senior residents the first 6 months of residency

Control group - gets the hospital's usual training and will receive the Bootcamp training starting at 6-month of residency.

The main thing the researchers want to know is: Does using the Boot Camp lower burnout-especially emotional exhaustion-compared with usual training? They will also look at the PHQ-9 depression survey and how confident residents feel about four everyday skills: mental health self-care, time management, oral presentation, and medical documentation. Surveys are completed at the start of residency and again six months later. Findings will show whether giving residents structured, on-demand preparation improves their well-being and confidence during the toughest part of their training.

DETAILED DESCRIPTION:
New interns often describe their first months of residency as a "trial by fire." Studies show that roughly one-third of U.S. residents develop significant depressive symptoms during training, and burnout-particularly feeling emotionally drained-has been linked to more medical errors and even suicidal thinking . OnlineMedEd's Intern Boot Camp (OME-IBC) is an on-demand video course endorsed by the American College of Physicians to help graduating medical students get ready for residency, yet no one has formally tested whether it actually improves interns' well-being in a busy urban hospital setting .

This single-center pilot study will recruit the entire 2024-2025 class of first-year residents at Harlem Hospital. After obtaining consent, participants complete a baseline survey and are then randomly assigned (1:1) to one of two groups, stratified by sex, specialty and Emotional Exhaustion score.

Intervention group - receives six months of free access to the password-protected OME-IBC website plus twice-weekly, one-hour review sessions led by senior residents. Each two- to three-week mini-unit focuses on one of four practical domains-mental-health self-care, time management, oral presentation, and documentation. Participants watch a short video together and discuss it. The full curriculum spans about 35 sessions and can also be viewed asynchronously.

Control group - follows the program's usual orientation and on-the-job teaching without Bootcamp access during the first six months. After the 6-month, they are offered the same OME-IBC access and review sessions.

Outcomes

Primary outcome: change in emotional-exhaustion scores on the Maslach Burnout Inventory (MBI). A ≥27 on the EE subscale indicates high burnout; every one-point rise has been tied to a 5-7 % jump in suicidal ideation or major errors.

Secondary outcomes:

Changes in overall burnout (other MBI subscales)

Depressive-symptom severity on the PHQ-9 (0-27 scale)

Self-rated confidence (1 = "minimally confident" to 5 = "very confident") in the four Bootcamp skill areas

ELIGIBILITY:
Inclusion Criteria:

* Incoming first year of residency

Exclusion Criteria:

* Previous United States Accredited Postgraduate Training
* PHQ-9 score above 20
* PHQ-9 positive for suicidality (question 9)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Burnout at 3 months and 6 months | Baseline measurement, post-intervention measurements at 3 months and 6 months
  The Maslach's burnout inventory is a 22-item measurement of worker burnout which assesses emotional exhaustion (EE), depersonalization (DP), and personal fulfillment (PF) domains. Possible scores range from 0-6 on a Likert scale for each item. Scores of EE ≥ 27 points, DP ≥ 10, and PF <33 would indicate a high degree of burnout. Scores of EE≤18 points, DP≤5 points, and PF≥40 points would indicate a low degree of burnout.

SECONDARY OUTCOMES:
Proportion of participants whose PHQ-9 total score is ≥ 10 at 3 months and 6 months | Baseline measurement, post-intervention measurements at 3 months and 6 months
  The Patient Health Questionnaire 9-item version (PHQ-9) to assess depressive symptoms. On PHQ-9, depression is categorized as minimal by a score of 0 to 4, mild by a score of 5 to 9, moderate by a score of 10 to 14, moderately severe by a score of 15 to 19, and severe by a score of 20 to 27. A total score ≥ 10 indicates clinically significant depressive symptoms. The outcome is the proportion of participants with a score ≥ 10 at 6 months. Lower proportions reflect better mental-health status.

CONTACTS AND LOCATIONS:
Overall Officials: Raji Ayinla, M.D., CMD, FCCP, FACP, Principal Investigator — New York City Health and Hospitals Corporation
Locations (1):
- Harlem Hospital Center, Manhattan, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the primary and secondary outcome results (baseline demographic variables, intervention allocation, PHQ-9, MBI, Mini-ReZ scores at baseline, 3 months and 6 months plus the data dictionary and statistical analysis code will be shared. Direct identifiers (name, email, MRN, full dates of birth) and high-risk elements (audio/video files, free-text survey comments) will not be shared to protect confidentiality in this small cohort.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 12 months after publication of the main results and for 5 years via the controlled-access repository Vivli
Access Criteria: Researchers with a methodologically sound proposal, IRB/ethics approval, and a signed data-use agreement may request access through the Vivli platform's review committee.

REFERENCES:
- [Background] Guille C, Zhao Z, Krystal J, Nichols B, Brady K, Sen S. Web-Based Cognitive Behavioral Therapy Intervention for the Prevention of Suicidal Ideation in Medical Interns: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Dec;72(12):1192-8. doi: 10.1001/jamapsychiatry.2015.1880. PMID 26535958